CLINICAL TRIAL: NCT01757457
Title: Anti-inflammatory Effects of Intracoronary and Intravenous Abciximab Administration During Primary Percutaneous Coronary Intervention.(Molecole di Adesione Nella Sindrome Coronarica Acuta
Brief Title: Anti-inflammatory Effects of Intracoronary and Intravenous Abciximab Administration During Primary Percutaneous Coronary Intervention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Lupi Alessandro, Principal Investigator, Azienda Ospedaliero Universitaria Maggiore della Carita
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0000004
Record Dates: First submitted 2012-12-19; First posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Myocardial Infarction
Keywords: inflammation; thrombosis; platelets; adhesion molecules; endothelium
MeSH Terms: conditions — Myocardial Infarction; Inflammation; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intracoronary abciximab (Experimental): Intracoronary administration of an abciximab bolus during primary PCI
  Interventions: Drug: Intracoronary administration of an abciximab bolus during primary PCI
- Intravenous abciximab (Active Comparator): Intravenous standard administration of an abciximab bolus during primary PCI
  Interventions: Drug: Intravenous administration of an abciximab bolus during primary PCI

INTERVENTIONS:
Drug: Intracoronary administration of an abciximab bolus during primary PCI — Intracoronary administration of an abciximab bolus (reopro 0.25mg/kg) during primary PCI
  Arms: Intracoronary abciximab
Drug: Intravenous administration of an abciximab bolus during primary PCI — Intracoronary administration of an abciximab bolus (reopro 0.25mg/kg) during primary PCI
  Arms: Intravenous abciximab

SUMMARY:
Intracoronary abciximab administration during primary percutaneous coronary intervention (pPCI) could offer clinical advantages over the intravenous route. The aim of this study was to assess whether abciximab administration route could influence its anti-inflammatory effects. 87 consecutive STEMI patients candidate to pPCI were randomized to receive an intracoronary or intravenous abciximab bolus. The primary endpoint was the extent of inflammation, measured by C-reactive protein (CRP), VCAM-1 and ICAM-1 levels.

DETAILED DESCRIPTION:
BACKGROUND: intracoronary abciximab administration during primary percutaneous coronary intervention (pPCI) could offer clinical advantages over the intravenous route. Besides antiplatelet effects, abciximab can modulate inflammation via cross-reactivity with GPIIb/IIIa, avb3, and aMb2 receptors. The aim of this study was to assess whether abciximab administration route could influence its anti-inflammatory effects.

METHODS: 87 consecutive STEMI patients candidate to pPCI were randomized to receive intracoronary (Group A, 47 patients) or intravenous (Group B, 42 patients) abciximab bolus. The primary endpoint was the extent of inflammation, measured by C-reactive protein (CRP), VCAM-1 and ICAM-1 levels.

ELIGIBILITY:
Inclusion Criteria:

* presence of STEMI according to the universal definition of myocardial infarction (7);
* hospital admission within 12 hours from symptom onset;
* successful treatment by primary PCI, defined as a procedure achieving infarct-related artery (IRA) patency with less than 10% residual coronary stenosis based on visual estimation.

Exclusion Criteria:

* age > 90 years;
* cardiogenic shock at admission;
* left main as IRA;
* saphenous vein graft as IRA;
* previous PCI in the last 6 months;
* severe renal impairment (eGFR<30ml/min) or dialysis treatment;
* thrombolytic drug administration in the last 30 days before admission;
* known malignancy diagnosed less than 5 years before admission;
* known active infectious, coagulative or systemic inflammatory diseases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Change in C-reactive protein levels from baseline after PCI | 48h
  C-reactive protein will be evaluated at admission and 48 hours after the primary PCI as marker of the inflammatory reaction

SECONDARY OUTCOMES:
Overall Mortality | 1year
  Mortality for all causes at 1year after primary PCI
Target vessel revascularization | 1 year
  Target vessel revascularization at 1 year after primary PCI
Myocardial infarction | 1 year
  Recurrent Myocardial infarction 1 year after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Lupi, MD, Principal Investigator — AO Maggiore della Carita
Locations (1):
- Ospedale Maggiore della Carità, Novara, Piedmont, Italy

REFERENCES:
- [Derived] Secco GG, Sansa M, Rognoni A, Parisi R, Fattori R, Rossi L, Lazzero M, Rolla R, Bellomo G, Bongo AS, Agostoni P, Di Mario C, Lupi A. Similar anti-inflammatory effects of intracoronary and intravenous abciximab during primary percutaneous coronary intervention: a randomized study. J Cardiovasc Med (Hagerstown). 2015 Mar;16(3):189-96. doi: 10.2459/JCM.0000000000000119. PMID 25022932